CLINICAL TRIAL: NCT04960709
Title: A Phase III Randomized, Open-Label, Multicenter Study to Determine the Efficacy and Safety of Durvalumab in Combination With Tremelimumab and Enfortumab Vedotin or Durvalumab in Combination With Enfortumab Vedotin for Perioperative Treatment in Patients Ineligible for Cisplatin or Who Refuse Cisplatin Undergoing Radical Cystectomy for Muscle Invasive Bladder Cancer (VOLGA)
Brief Title: Treatment Combination of Durvalumab, Tremelimumab and Enfortumab Vedotin or Durvalumab and Enfortumab Vedotin in Patients With Muscle Invasive Bladder Cancer Ineligible to Cisplatin or Who Refuse Cisplatin
Acronym: VOLGA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D910PC00001; 2020-005452-38 (EudraCT Number)
Record Dates: First submitted 2021-06-17; First posted 2021-07-14 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Muscle Invasive Bladder Cancer
Keywords: Bladder Cancer; Immunotherapy; PD-L1; Durvalumab (MEDI4736); Tremelimumab; Enfortumab Vedotin (PADCEV)
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — durvalumab; tremelimumab; enfortumab vedotin; Cystectomy

STUDY DESIGN:
Intervention Model Description: Parallel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Durvalumab + Tremelimumab + Enfortumab Vedotin (Experimental): Participants will receive 3 preoperative 21-day cycles of Durvalumab + Enfortumab Vedotin and 2 cycles of Tremelimumab, followed by radical cystectomy, followed by 1 cycle of postoperative Tremelimumab and 9 cycles of Durvalumab. Each postoperative cycle is 28 days.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Enfortumab Vedotin; Procedure: Radical Cystectomy
- Durvalumab + Enfortumab vedotin (Experimental): Participants will receive 3 preoperative 21-day cycles of Durvalumab + Enfortumab Vedotin, followed by radical cystectomy, followed by 9 cycles of Durvalumab. Each postoperative cycle is 28 days.
  Interventions: Drug: Durvalumab; Drug: Enfortumab Vedotin; Procedure: Radical Cystectomy
- Cystectomy with or without approved Adjuvant Therapy. (Active Comparator): Participants may receive SoC (nivolumab approved as adjuvant treatment for MIBC based on high risk criteria) per approved label in the country OR Participants receive standard of care surgery (radical cystectomy) alone.
  Interventions: Procedure: Radical Cystectomy

INTERVENTIONS:
Drug: Durvalumab — Anti- PD-L1 Antibody
  Other Names: IMFINZI; MEDI4736
  Arms: Durvalumab + Enfortumab vedotin; Durvalumab + Tremelimumab + Enfortumab Vedotin
Drug: Tremelimumab — Human IgG2 mAb
  Arms: Durvalumab + Tremelimumab + Enfortumab Vedotin
Drug: Enfortumab Vedotin — Nectin-4-directed antibody and microtubule inhibitor conjugate
  Other Names: PADCEV
  Arms: Durvalumab + Enfortumab vedotin; Durvalumab + Tremelimumab + Enfortumab Vedotin
Procedure: Radical Cystectomy — For cisplatin-ineligible or cisplatin-refusal patients

SUMMARY:
A global phase 3, multicenter, randomized, trial, to Determine the Efficacy and Safety of Durvalumab in combination with Tremelimumab and Enfortumab Vedotin or Durvalumab in combination with Enfortumab Vedotin for Perioperative Treatment in Patients Ineligible for Cisplatin or who refuse Cisplatin based chemotherapy Undergoing Radical Cystectomy for Muscle Invasive Bladder Cancer.

The goal of the study is to explore the triplet combination of Durvalumab, Tremelimumab and Enfortumab Vedotin or the duplet combination of Durvalumab and Enfortumab vedotin in terms of efficacy and safety compared to the current Standard Of Care (SOC).

VOLGA trial consists of two parts: Safety Run-In and Main Study. In total the study aims to enroll approximately 677 patients, who will receive triplet combination, duplet combination or currently approved SOC in the main study. In the main part of the trial there is two out of three chances of being on a treatment arm and the treatment is assigned at random by a computer system.

In this trial patients in the two treatment arms will receive either 3 cycles of neoadjuvant Durvalumab + Enfortumab Vedotin and 2 cycles of Tremelimumab or Durvalumab + Enfortumab vedotin and after surgery both treatment arms will receive either adjuvant Durvalumab or adjuvant Durvalumab and 1 cycle of Tremelimumab.

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented muscle-invasive UC of the bladder.
* Participants with transitional cell and mixed transitional/non-transitional cell histologies;
* Participants with MIBC clinical tumor (T) stage T2-T4aN0/1M0 or UC of the bladder with clinical state T1N1M0 (participants with T1 stage are allowed only with N1 disease)
* Participants should also have not received prior systemic chemotherapy or immunotherapy for the treatment of MIBC or bladder UC.
* Medically fit for cystectomy and able to receive neoadjuvant therapy;
* Patients who have not received prior systemic chemotherapy or immunotherapy for treatment of MIBC;
* ECOG performance status of 0,1,2 at enrollment.
* Availability of tumor sample prior to study entry;
* Must have a life expectancy of at least 12 weeks at randomization.
* Cisplatin-ineligible, following criteria based on Galsky et al 2011 OR Refuse cisplatin based chemotherapy (must be documented in the medical records)

Exclusion criteria:

* Evidence of lymph node (N2+) or metastatic TCC/UC disease at the time of screening.
* Active infection
* Uncontrolled intercurrent illness
* Prior exposure to immune-mediated therapy (with exclusion of Bacillus-Calmette Guerin [BCG]), including but not limited to other anti-CTLA-4, anti--PD-1, anti PD-L1, or anti-PD-L2 antibodies.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of IPs.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-09-08 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability as evaluated by adverse events occurring throughout the study (Safety Run-In part) | At completion of study treatment by the last patient and at 3 months.
  Frequency of Adverse Events.
To assess the safety and tolerability of durvalumab + tremelimumab + EV in participants with MIBC who are ineligible for cisplatin as assessed by vital signs (blood pressure in mmHg) (Safety Run-In part) | Up to 84 months
To assess the safety and tolerability of durvalumab + tremelimumab + EV in participants with MIBC who are ineligible for cisplatin as assessed by vital signs (pulse rate) in beats per minute (Safety Run-In part) | Up to 84 months
To assess the safety and tolerability of durvalumab + tremelimumab + EV in participants with MIBC who are ineligible for cisplatin as assessed by vital signs (respiration rate) in breaths per minute (Safety Run-In part) | Up to 84 months
To assess the safety and tolerability of durvalumab + tremelimumab + EV in participants with MIBC who are ineligible for cisplatin as assessed by vital signs (temperature) in degrees Celsius (Safety Run-In part) | Up to 84 months
To assess the safety and tolerability of durvalumab + tremelimumab + EV in participants with MIBC who are ineligible for cisplatin as assessed by abnormality in clinical chemistry by liver function (Safety Run-In part) | Up to 84 months
  Clinical chemistry will be assessed by liver function assessment (ALT, AST, albumin, total bilirubin measured in units per dL)
Safety and tolerability of durvalumab + tremelimumab + EV in participants with MIBC who are ineligible for cisplatin or who refuse cisplatin as assessed by abnormality in clinical chemistry by kidney function (Safety Run-In part) | Up to 84 months
  Clinical chemistry will be assessed by kidney function assessment in mg/dL
To assess the safety and tolerability of durvalumab + tremelimumab + EV in participants with MIBC who are ineligible for cisplatin as assessed by abnormality in clinical chemistry by thyroid function (Safety Run-In part) | Up to 84 months
  Clinical chemistry will be assessed by thyroid function assessment in units per mL.
To assess the safety and tolerability of durvalumab + tremelimumab + EV in participants with MIBC who are ineligible for cisplatin as assessed by abnormality in haematology (Safety Run-In part) | Up to 84 months
  Hematology will be assessed by white cell count, platelet count, absolute neutrophil count and absolute lymphocyte count.
To assess the safety and tolerability of durvalumab + tremelimumab + EV in participants with MIBC who are ineligible for cisplatin as as assessed by ECG (pulse rate) (Safety Run-In part) | Up to 84 months
Changes in WHO/ECOG performance status (Safety Run-In part) | Up to 84 months
  Eastern Cooperative Oncology Group (ECOG) performance status scale range 0 to 5, where 0 is fully active, able to carry on all pre disease performance without restriction - best outcome and 5 -death - worst outcome.
Compare efficacy of durvalumab + tremelimumab + EV (Arm 1) relative to cystectomy (Arm 3) and durvalumab + EV (Arm 2) relative to cystectomy (Arm 3) on EFS (Main Study) | Up to 3 years
  Event-free survival (EFS;) is defined as the time from randomization to the first occurrence of any of the following events: recurrence of disease post-radical cystectomy, the first documented progression in participants who did not receive radical cystectomy, failure to undergo radical cystectomy in participants with residual disease, or death due to any cause, up to 3 years.

SECONDARY OUTCOMES:
1. To evaluate the efficacy of durvalumab + tremelimumab + EV on pCR rate (Safety Run-in part) | 3 years
  Pathologic complete response (pCR) rate is defined as the number of participants whose pathological staging was T0N0M0 as assessed per local pathology and central independent review using specimens obtained via cystectomy, at 3 years.
2. To evaluate the efficacy of durvalumab + tremelimumab + EV on EFS (Safety Run-in part) | 3 years
  Event-free survival (EFS;) is defined as the time from randomization to the first occurrence of any of the following events: recurrence of disease post-radical cystectomy, the first documented progression in participants who did not receive radical cystectomy, failure to undergo radical cystectomy in participants with residual disease, or death due to any cause, up to 3 years.
3. Pathologic complete response (pCR) rates at time of cystectomy in Arm1 vs Arm3 and Arm 2 vs Arm 3 (Main Study part) | 3 years
  Pathologic complete response (pCR) rate is defined as the number of participants whose pathological staging was T0N0M0 as assessed per local pathological review using specimens obtained via cystectomy, at 3 years.
4. Overall survival (Safety Run-in and Main Study part) | Up to 5 years
  Overall Survival is defined as length of time from randomization until the date of death due to any cause, whichever came first, assessed up to 5 years.
5. EFS at 24 months (EFS24) (Safety Run-in and Main Study part) | Up to 24 months
  EFS24 is defined as proportion of participants alive and event-free at 24 months
6. Overall survival rate at 5 years (Safety Run-in and Main Study part) | At 5 years
  The proportion of participants alive at 5 years (OS5) is defined as the Kaplan-Meier estimate of OS at 5 years after randomization
7. Disease-free survival (DFS) (Safety Run-in and Main Study part) | Up to first recurrence of disease or death up to 5 years
  DFS is defined as time from radical cystectomy to recurrence or death, whichever came first, assessed up to 5 years.
8. Pathologic downstaging (pDS) rate-to < pT2 (Safety Run-in and Main Study part) | 3 years
  pDS rate is defined as the rate of downstaging to < pT2, including pT0, pTis, pTa, pT1, and N0
9. Disease-specific survival (DSS) (Safety Run-in and Main Study part) | from randomization until death due to bladder cancer up to 5 year.
  DSS is defined as time from randomization until death due to bladder cancer, assessed up to 5 years.
10. EORTC QLQ-C30 European Organisation for Research and Treatment of Cancer 30-item Core Quality of Life Questionnaire) (Safety Run-in and Main Study part) | from baseline and time to definitive clinically, assessed up to 5 years
11. Immunogenicity of durvalumab when used in combination with Tremelimumab as measured by presence of antidrug antibodies (ADA) (Safety Run-in and Main Study part) | At 3 months after last dose of durvalumab and tremelimumab
12. Time to maximum observed serum concentration (tmax) of durvalumab and tremelimumab (Safety Run-in and Main Study part) | At 3 months after last dose of durvalumab and tremelimumab
13. Metastasis-free survival (MFS) (Safety Run-in and Main Study part) | From randomization until the first recognition of distant metastases or death, up to approximately 48 months.
  MFS is defined as the time from date of randomization until the first recognition of distant metastases or death, whichever occurs first, up to approximately 48 months.

CONTACTS AND LOCATIONS:
Locations (168):
- United States (31):
  - Research Site, Orange, California
  - Research Site, Santa Monica, California
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fort Myers, Florida
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Maywood, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, Scarborough, Maine
  - Research Site, Boston, Massachusetts
  - Research Site, Brighton, Michigan
  - Research Site, Jackson, Mississippi
  - Research Site, Las Vegas, Nevada
  - Research Site, Saddle Brook, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Syracuse, New York
  - Research Site, Portland, Oregon
  - Research Site, Hershey, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Knoxville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Spokane, Washington
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Pergamino
  - Research Site, Pilar
- Austria (6):
  - Research Site, Graz
  - Research Site, Krems
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Wiener Neustadt
- Brazil (10):
  - Research Site, Barretos
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santa Maria
  - Research Site, Santo André
  - Research Site, São Paulo
  - Research Site, Săo Paulo
  - Research Site, Uberlândia
- Canada (4):
  - Research Site, Abbotsford, British Columbia
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- Research Site, Santiago, Chile
- France (14):
  - Research Site, Amiens
  - Research Site, Bayonne
  - Research Site, Clermont-Ferrand
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Pierre-Bénite
  - Research Site, Quint-Fonsegrives
  - Research Site, Saint-Priez En Jarez
  - Research Site, Strasbourg
  - Research Site, Suresnes
  - Research Site, Vandœuvre-lès-Nancy
- Germany (15):
  - Research Site, Bielefeld
  - Research Site, Bochum
  - Research Site, Cologne
  - Research Site, Düsseldorf
  - Research Site, Giessen
  - Research Site, Hanover
  - Research Site, Herne
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Münster
  - Research Site, Regensburg
  - Research Site, Reutlingen
  - Research Site, Ulm
- Greece (2):
  - Research Site, Athens
  - Research Site, Maroussi, Athens
- Research Site, Shatin, Hong Kong
- Israel (4):
  - Research Site, Hadera
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Tel Aviv
- Italy (11):
  - Research Site, Bari
  - Research Site, Florence
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Pozzuoli
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Terni
  - Research Site, Tricase
  - Research Site, Verona
- Japan (19):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hamamatsu
  - Research Site, Ichikawa-shi
  - Research Site, Kanazawa
  - Research Site, Kashihara-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kita-gun
  - Research Site, Kobe
  - Research Site, Kumamoto
  - Research Site, Matsuyama
  - Research Site, Miyazaki
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Toyama
  - Research Site, Tsukuba
  - Research Site, Yokohama
- Mexico (2):
  - Research Site, Colima
  - Research Site, Monterrey
- Netherlands (6):
  - Research Site, Arnhem
  - Research Site, Breda
  - Research Site, Groningen
  - Research Site, Hoofddorp
  - Research Site, Leiden
  - Research Site, Utrecht
- Poland (4):
  - Research Site, Gdansk
  - Research Site, Nowa Sól
  - Research Site, Skórzewo
  - Research Site, Warsaw
- Portugal (4):
  - Research Site, Braga
  - Research Site, Coimbra
  - Research Site, Faro
  - Research Site, Lisbon
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Kamenitz
- South Korea (5):
  - Research Site, Busan
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (6):
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Seville
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Tainan
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Dusit
  - Research Site, Songkhla
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Karşıyaka
- Research Site, London, United Kingdom
- Vietnam (4):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Huế

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home